CLINICAL TRIAL: NCT05359380
Title: Evaluation of the Impact of Light Intensity and Light Temperature on the Efficacy of Presbyopic Corrections With Bilateral Implantation of Multifocal Intraocular Lenses in a Series of Activities of Daily Living
Brief Title: The Impact of Light Conditions on the Efficacy of Multifocal Intraocular Lens Implantation in Activities of Daily Living
Status: Completed | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES1/Th1/08-02-2018
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Presbyopia; Near Vision; Reading; Daily Activities; Multifocal Intraocular Lens; Cataract
Keywords: activities of daily living; presbyopia; light temperature; light intensity; multifocal intraocular lens
MeSH Terms: conditions — Presbyopia; Myopia; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SG1 - Trifocal Group: Patients implanted bilaterally with trifocal diffractive IOLs
  Interventions: Other: ADL performance
- SG2 - Bifocal Group: Patients implanted bilaterally with bifocal hybrid (diffractive - refractive) IOLs
  Interventions: Other: ADL performance
- SG3 - Monofocal Group: Patients implanted bilaterally with monofocal IOLs
  Interventions: Other: ADL performance

INTERVENTIONS:
Other: ADL performance — ADL performance
  All study groups address the following 10 ADL tasks in 9 different combinations of light temperature and light intensity in order possible differences to be revealed among the study groups and light combinations:
  1. Phone Book Search (PBS), 2. Supermarket receipt (SupRe), 3. Book reading (BR), 4. Cellular message (CM), 5. Cellular entry search (CES), 6. Reading computer screen (RCS), 7. Drops bottle reading (DR), 8. Subtitles reading (SubRe), 9. Open door test (ODT), and, 10. Screwdriver test (ST).
  The 9 light combinations are the following:
  3000 K - 25 fc, 3000 K - 50 fc, 3000 K - 75 fc / 4000 K - 25 fc, 4000 K - 50 fc, 4000 K - 75 fc / 6000 K - 25 fc, 6000 K - 50 fc, 6000 K - 75 fc

SUMMARY:
Primary objective of this study is to identify the optimal task lighting conditions (in terms of light intensity and light temperature) for 10 activities of daily living (ADLs) that require near or intermediate vision acuity in a validated ADL simulation framework for a sample of patients who underwent presbyopic correction with bilateral multifocal intraocular lenses (IOLs) implantation, and to compare their capacity to perform ADLs (ADL scores) between three study groups (SG): SG1. patients implanted bilaterally with trifocal diffractive IOLs, SG2. patients implanted bilaterally with bifocal hybrid (diffractive-refractive) IOLs, SG3. patients implanted bilaterally with monofocal IOLs

DETAILED DESCRIPTION:
Patients who underwent presbyopic correction with bilateral implantation of multifocal IOLs are supposed to have sufficient uncorrected vision capacity for ADLs that require near (ie. book reading) or intermediate (ie. reading in a computer screen) vision acuity. However, it is known that light intensity and light temperature has a great impact on near/intermediate vision capacity, but also patients that have been implanted with multifocal IOLs are most likely to present completely different lighting needs than patients with their own crystalline lenses.

Primary objective of this study is to identify the optimal task lighting conditions (in terms of light intensity and light temperature) for 10 ADLs that require near or intermediate vision acuity in a validated ADL simulation framework for a sample of patients who underwent presbyopic correction with bilateral multifocal IOLs implantation, and to compare their capacity to perform the ADLs (ADL scores) in 9 different lighting combinations (combinations of light intensity and light temperature) between three study groups: SG1. patients implanted bilaterally with trifocal diffractive IOLs, SG2. patients implanted bilaterally with bifocal hybrid (diffractive-refractive) IOLs, SG3. patients implanted bilaterally with monofocal IOLs

The study is conducted in an experimental facility in a hospital room with a dimension of 6.87 × 2.9 × 3 m (depth × width × height) and flat white surface walls (reflectance: 70%). Αn advanced light diffusion system has been installed, which consists of four linear LED luminaires producing low glare (unified glare rating (UGR) < 19). Light intensity (dimming / in foot candles - fc) and light temperature (white tuning / (in Kelvins - K) have been adjusted using the Casambi wireless control application (Casambi Technologies Oy Inc., Espoo, Finland), which uses integrated Bluetooth mesh technology and secures maximal uniformity at different user-defined lighting settings. The four LED luminaires have been mounted on the ceiling. The exact luminaire positioning and the amount of the provided luminous flux have been defined using the RELUX light simulation tool (version 2021.1.1.0) (Relux Informatik AG, Münchenstein, Switzerland) prior to the installation. The confirmation of illuminance and on-site adjustments have been confirmed with the Extech Lux Meter EA30 (Extech Instruments Corporation, Nashua, NH, United States). As regards photometric properties derived from lighting laboratory photometric measurements, the correlated color temperature (CCT) of the luminaires ranges between 2700 K and 6500 K, emitting a maximum luminous flux of 10,626 lm and 11,508 lm, respectively. The exact radiant flux P(λ) emitted from the selected light sources has been measured using a Konica Minolta CL-500A spectrum meter for the wavelength range of 380-780 nm using a step of 1 nm. The power of each luminaire is 106 W, resulting in luminous efficacy of 100.2 lm/W and 108.6 lm/W for 2700 K and 6500 K, respectively. The color rendering index (CRI) is 84. The wireless dimming control system enables dimming from 0% to 100% and vice versa.

The 9 lighting combinations (light intensity, light temperature) are the following:

3000 K - 25 fc, 3000 K - 50 fc, 3000 K - 75 fc / 4000 K - 25 fc, 4000 K - 50 fc, 4000 K - 75 fc / 6000 K - 25 fc, 6000 K - 50 fc, 6000 K - 75 fc

In specific, patients address the following ten ADLs:

1. Phone Book Search (PBS), 2. Supermarket receipt (SupRe), 3. Book reading (BR), 4. Cellular message (CM), 5. Cellular entry search (CES), 6. Reading computer screen (RCS), 7. Drops bottle reading (DR), 8. Subtitles reading (SubRe), 9. Open door test (ODT), and, 10. Screwdriver test (ST).

Test-retest reliability will be assessed by calculating intraclass correlation coefficients (ICCs) for all ADLs at the nine combinations of light conditions in two different visits with an average 15-day time window to prevent memory effect.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years old
* Diagnosis of senile cataract either stage 2 or 3 of the Lens Opacities Classification System III (LOCS-3) grading scale - Patients underwent phacoemulsification and bilateral implantation of IOLs [trifocal diffractive, bifocal hybrid (diffractive - refractive) or monofocal]
* Fluency in written and verbal Greek language
* No severe cognitive impairment

Exclusion Criteria:

* Αstigmatism >1.00 diopters
* Glaucoma
* Intraocular pressure-lowering medications
* Corneal pathology
* Fundus pathology
* Diabetes mellitus
* Autoimmune diseases
* Former incisional eye surgery
* Posterior capsule rupture or lens misalignment
* Neurological, psychiatric or mental diseases that interfere with visual acuity and reading process
* Inability to understand the objectives of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent phacoemulsification and bilateral implantation of IOLs [SG1: trifocal diffractive IOL, SG2: bifocal hybrid (diffractive - refractive) IOL, SG3: monofocal IOL]
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Phone Book Search (PBS) score | through study completion, an average of 6 months
  Patient is required to find and read a specific entry in a regular phonebook catalog in the nine different combinations of light temperature and light intensity. A different entry is asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Supermarket Receipt (SupRe) score | through study completion, an average of 6 months
  Patient is required to find and read three products from a typical supermarket receipt in the nine different combinations of light temperature and light intensity. Different products are asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Book Reading (BR) score | through study completion, an average of 6 months
  Patient is required to read an excerpt of a predetermined length in a novel in the nine different combinations of light temperature and light intensity. A different excerpt of the same length is asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Cellular message (CM) score | through study completion, an average of 6 months
  Patient is required to read a Short Message Service (SMS) on a cellular phone in the nine different combinations of light temperature and light intensity. A different SMS is asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Cellular Entry Search (CES) score | through study completion, an average of 6 months
  Patient is required to find and read one specific entry on a cellular phone in the nine different combinations of light temperature and light intensity. Different entries are asked to be found in each combination.
  [scale's best value: 100, scale's worst value: 0]
Reading Computer Screen (RCS) score | through study completion, an average of 6 months
  Patient is required to correctly read text of a predetermined length from a computer screen in the nine different combinations of light temperature and light intensity. Different texts of the same length are asked to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Drops bottle Reading (DR) score | through study completion, an average of 6 months
  Patient is required to correctly read the expiration date printed on three typical eye dropper bottles in the nine different combinations of light temperature and light intensity. Different eye dropper bottles are given to be read in each combination.
  [scale's best value: 100, scale's worst value: 0]
Subtitles Reading (SubRe) score | through study completion, an average of 6 months
  Patient is required to correctly read movie subtitles from a one-minute movie excerpt on a computer screen in the nine different combinations of light temperature and light intensity. Different movie excerpts are shown in each combination.
  [scale's best value: 100, scale's worst value: 0]
Open Door Test (ODT) score | through study completion, an average of 6 months
  Patient is required to find a specific key from a keychain that holds 10 keys and put it in the corresponding door keyhole in the nine different combinations of light temperature and light intensity. Different keychains are given in each combination.
  [scale's best value: 100, scale's worst value: 0]
Screwdriver Test (ST) score | through study completion, an average of 6 months
  Patient is required to select one among three screwdrivers and insert it in the appropriate screw among a variety of screw types in the nine different combinations of light temperature and light intensity. Different screwdrivers are given to be selected in each combination.
  [scale's best value: 100, scale's worst value: 0]

SECONDARY OUTCOMES:
Uncorrected Distance Visual Acuity (UDVA) | through study completion, an average of 6 months
  Monocular and binocular UDVA of all groups is estimated using the Greek version of the Early Treatment Diabetic Retinopathy Study Chart at four meters distance
Uncorrected Intermediate Visual Acuity (UIVA) | through study completion, an average of 6 months
  Monocular and binocular UIVA of all groups is estimated using web-based Democritus Digital Acuity Reading Test (wDDART)
Uncorrected Near Visual Acuity (UNVA) | through study completion, an average of 6 months
  Monocular and binocular UNVA of all groups is estimated using web-based Democritus Digital Acuity Reading Test (wDDART)
25-item National Eye Institute Visual Function Questionnaire (NEI VFQ-25) score | through study completion, an average of 6 months
  Vision-specific quality of life of all participants is evaluated with the Greek version of NEI VFQ-25, which is handed to the patients prior to their ADL assessment.
Subjective preference of lighting combination | through study completion, an average of 6 months
  Patients are asked to choose the most preferable combination of light intensity and light temperature among the 9 different combinations for the most comfortable performance in ADLs

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, Study Chair — Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupolis, Greece
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

REFERENCES:
- [Background] Labiris G, Panagiotopoulou EK, Ntonti P. Development and Validation of a Lighting Facility for the Objective Assessment of the Visual Performance of Presbyopic Patients in a Series of Activities of Daily Living. Cureus. 2022 Apr 28;14(4):e24548. doi: 10.7759/cureus.24548. eCollection 2022 Apr. PMID 35651385
- [Background] Labiris G, Panagiotopoulou EK, Taliantzis S, Perente A, Delibasis K, Doulos LT. Lighting Standards Revisited: Introduction of a Mathematical Model for the Assessment of the Impact of Illuminance on Visual Acuity. Clin Ophthalmol. 2021 Nov 28;15:4553-4564. doi: 10.2147/OPTH.S326139. eCollection 2021. PMID 34866900
- [Background] Labiris G, Panagiotopoulou EK, Duzha E, Tzinava M, Perente A, Konstantinidis A, Delibasis K. Development and Validation of a Web-Based Reading Test for Normal and Low Vision Patients. Clin Ophthalmol. 2021 Sep 22;15:3915-3929. doi: 10.2147/OPTH.S314943. eCollection 2021. PMID 34588763